CLINICAL TRIAL: NCT04747977
Title: A Randomized, Double-Masked, Vehicle-Controlled, Phase 2 Study to Evaluate the Efficacy and Safety of OTX-DED (Dexamethasone Intracanalicular Ophthalmic Insert) for the Short-Term Treatment of Signs and Symptoms of Dry Eye Disease (DED)
Brief Title: To Assess the Efficacy and Safety of OTX-DED for the Short-term Treatment of Signs and Symptoms of Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTX-DED-2020-201
Record Dates: First submitted 2021-02-04; First posted 2021-02-10 (Actual); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: Dry Eye
Keywords: dexamethasone ophthalmic insert
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Parallel: Participants are assigned to one of two or more groups in parallel for the duration of the study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OTX-DED 0.2mg (Experimental): Approximately 50 subjects
  Interventions: Drug: OTX-DED
- OTX-DED 0.3mg (Experimental): Approximately 50 subjects
  Interventions: Drug: OTX-DED
- Hydrogel Vehicle (HV) (Placebo Comparator): Approximately 50 subjects
  Interventions: Drug: OTX-DED

INTERVENTIONS:
Drug: OTX-DED — 0.2mg dexamethasone ophthalmic insert
  Arms: OTX-DED 0.2mg
Drug: OTX-DED — 0.3mg dexamethasone ophthalmic insert
  Arms: OTX-DED 0.3mg
Drug: OTX-DED — Hydrogel vehicle ophthalmic insert
  Arms: Hydrogel Vehicle (HV)

SUMMARY:
To assess the efficacy and safety of OTX-DED for the short-term treatment of signs and symptoms of dry eye disease.

DETAILED DESCRIPTION:
Randomized, double-masked, vehicle-controlled, phase 2 study evaluating the efficacy and safety of OTX-DED (dexamethasone intracanalicular ophthalmic insert) for the short-term treatment of signs and symptoms of Dry Eye Disease (DED). The subjects will be followed for approximately 2-3 months from screening to the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Dry Eye Disease diagnosis
* VAS eye dryness severity score ≥ 40.

Exclusion Criteria:

* Are unwilling to discontinue use of contact lenses
* Are unwilling to withhold use of artificial tears.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-09-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Ocular Therapeutix, Inglewood, California
  - Ocular Therapeutix, Inc, Mission Hills, California
  - Ocular Therapeutix, Inc., Newport Beach, California
  - Ocular Therapeutix, Inc., Santa Ana, California
  - Ocular Therapeutix, Inc., Delray Beach, Florida
  - Ocular Therapeutix, Inc., Largo, Florida
  - Ocular Therapeutix, Warrenville, Illinois
  - Ocular Therapeutix, Inc., Indianapolis, Indiana
  - Ocular Therapeutix, Kansas City, Missouri
  - Ocular Therapeutix, Inc., St Louis, Missouri
  - Ocular Therapeutix, Poughkeepsie, New York
  - Ocular Therapeutix, Inc., Raleigh, North Carolina
  - Ocular Therapeutix, Inc., Cranberry Township, Pennsylvania
  - Ocular Therapeutix, Inc., Memphis, Tennessee
  - Ocular Therapeutix, Inc., League City, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- OTX-DED 0.2mg Dexamethasone Intracanalicular Ophthalmic Insert: Subjects in this arm received 0.2mg Dexamethasone Intracanalicular Ophthalmic Insert
- OTX-DED 0.3mg Dexamethasone Intracanalicular Ophthalmic Insert: Subjects in this arm received 0.3mg Dexamethasone Intracanalicular Ophthalmic Insert
- Hydrogel Vehicle (HV) Intracanalicular Insert: Subjects in this arm received Hydrogel Vehicle (HV) Intracanalicular Insert
Period: Overall Study
Arm/Group | OTX-DED 0.2mg Dexamethasone Intracanalicular Ophthalmic Insert | OTX-DED 0.3mg Dexamethasone Intracanalicular Ophthalmic Insert | Hydrogel Vehicle (HV) Intracanalicular Insert
Started | 57 | 57 | 58
Completed | 54 | 56 | 55
Not Completed | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Population: The Modified Intent-to-Treat (mITT) analysis set includes all subjects in the Intent-to-Treat (ITT) population who received IP (OTX-DED or HV) in the study eye.
Groups:
- Total: Total of all reporting groups
Arm/Group | OTX-DED 0.2mg Dexamethasone Intracanalicular Ophthalmic Insert | OTX-DED 0.3mg Dexamethasone Intracanalicular Ophthalmic Insert | Hydrogel Vehicle (HV) Intracanalicular Insert | Total
Number analyzed (Participants) | 55 | 56 | 55 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (11.0) | 65.4 (11.4) | 63.8 (12.3) | 64.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 39 | 41 | 121
  Male | 14 | 17 | 14 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 4 | 6 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 14 | 8 | 33
  White | 39 | 38 | 41 | 118
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Photographic Assessment of Bulbar Conjunctival Hyperemia Change in Score From Baseline (CFB) at 15 Days (Evaluated Via Central Reading Center).
Description: The primary efficacy endpoint is photographic assessment of bulbar conjunctival hyperemia [evaluated by the central reading center (CRC)] in the study eye, change in score from baseline (CFB) at Visit 4 (Day 15).
  Scoring is from 0 (None) to 4 (Severe) on the CCLRU Grading Scale for Bulbar Conjunctival Hyperemia.
Time Frame: Change from baseline (Day 1) at Visit 4 (Day 15)
Population: mITT population: CFB in Photographic Assessment of Bulbar Conjunctival Hyperemia in the Worst Zone (highest grading score at baseline among nasal, temporal, and frontal zones) of Study Eye at Day 15
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | OTX-DED 0.2mg Dexamethasone Intracanalicular Ophthalmic Insert | OTX-DED 0.3mg Dexamethasone Intracanalicular Ophthalmic Insert | Hydrogel Vehicle (HV) Intracanalicular Insert
Number analyzed (Participants) | 55 | 56 | 55
score on a scale | -0.51 [-0.65 to -0.37] | -0.43 [-0.57 to -0.30] | -0.21 [-0.35 to -0.07]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 10 weeks.
Description: This analysis includes the Modified Intent To Treat (mITT) analysis set which includes all subjects in the Intent To Treat (ITT) population who received IP (OTX-DED or HV) in the study eye.
Arm/Group | OTX-DED 0.2mg Dexamethasone Intracanalicular Ophthalmic Insert | OTX-DED 0.3mg Dexamethasone Intracanalicular Ophthalmic Insert | Hydrogel Vehicle (HV) Intracanalicular Insert
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/56 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56 | 2/55
Other Adverse Events (participants affected / at risk) | 5/55 | 10/56 | 6/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OTX-DED 0.2mg Dexamethasone Intracanalicular Ophthalmic Insert (N=55) | OTX-DED 0.3mg Dexamethasone Intracanalicular Ophthalmic Insert (N=56) | Hydrogel Vehicle (HV) Intracanalicular Insert (N=55)
Cellulitis/Worsening of Cellulitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OTX-DED 0.2mg Dexamethasone Intracanalicular Ophthalmic Insert (N=55) | OTX-DED 0.3mg Dexamethasone Intracanalicular Ophthalmic Insert (N=56) | Hydrogel Vehicle (HV) Intracanalicular Insert (N=55)
Eye Disorders (Eye disorders) | 5 | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT04747977/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT04747977/SAP_001.pdf